CLINICAL TRIAL: NCT07311161
Title: The Efficacy of Dysphagia Digital Therapy in Patients With Various Swallowing Disorders: A Pilot Study
Brief Title: Dysphagia Digital Therapy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024-03-005
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia Rehabilitation
Keywords: mobile application; digital therapeutics

STUDY DESIGN:
Intervention Model Description: This was a single-center, prospective, case series pilot study. Participants were diagnosed as dysphagia after VFSS.
  Two sessions of swallowing therapy and digital therapeutic (DTx) education were conducted by an occupational therapist to familiarize the participant. Each participant then performed individualized home-based swallowing exercises using the DTx application for 4 weeks, three times daily.
  The individuals allowed a preliminary evaluation of the feasibility and applicability of the mobile-based digital therapeutic intervention across a broad spectrum of dysphagia etiologies.
  The primary outcome of this study was the assessment of airway protection using the Penetration-Aspiration Scale (PAS) evaluated through videofluoroscopic swallowing study (VFSS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with dysphagia (Experimental)
  Interventions: Device: "Pallow", mobile-based digital therapeutic (DTx)

INTERVENTIONS:
Device: "Pallow", mobile-based digital therapeutic (DTx) — mobile-based digital therapeutic (DTx) application designed for swallowing rehabilitation

SUMMARY:
Dysphagia is a swallowing disorder characterized by impaired transfer of food or liquid from the oral cavity through the pharynx and esophagus, leading to significant nutritional, respiratory, and quality-of-life consequences.

Despite these advances, existing dysphagia rehabilitation programs are largely limited to specific disease groups, restricting their generalizability. In clinical practice, dysphagia arises from diverse etiologies, including stroke, neurodegenerative diseases, and other neurological or muscular conditions, which share common rehabilitation goals such as safe swallowing, aspiration prevention, and maintenance of oral intake.

This pilot study aimed to evaluate the feasibility and preliminary effectiveness of a novel mobile-based digital therapeutic (DTx) application for dysphagia rehabilitation across a clinically heterogeneous population. The DTx platform leverages mobile device camera signals to provide real-time feedback, structured reminders, and quantitative monitoring of self-directed training. We hypothesized that integrating this DTx into dysphagia care would enhance patient engagement, adherence, and swallowing-related outcomes. The findings of this study are expected to inform future large-scale trials and support the broader implementation of digital therapeutics in dysphagia rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years with dysphagia from head and neck cancer surgery/chemotherapy, cerebrovascular/neurodegenerative diseases, or neuromuscular diseases
2. Swallowing difficulty, indicated by Penetration-Aspiration Score (PAS) ≥2 by VFSS
3. Ability to sit for more than 30 minutes
4. no significant cognitive impairment and mobile device access (MMSE>24)

Exclusion Criteria:

1. Participants who need hospitalization (e.g. pneumonia)
2. Requirement of surgical treatment during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale (PAS) | From enrollment to the end of intervention at 4 weeks
  Penetration and aspiration are evaluated using an 8-point scale during a Videofluoroscopic Swallowing Study (VFSS) to determine the severity of airway invasion. Scores range from 1 (normal) to 8 (material passes below the vocal folds with no effort to eject). The higher the score, the more severe the dysphagia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea